CLINICAL TRIAL: NCT05884359
Title: Left Bundle Branch Area Mapping for Conduction System Pacing
Status: Recruiting | Type: Observational
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: SEMC
Record Dates: First submitted 2023-04-18; First posted 2023-06-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Left Bundle-Branch Block; Pacemaker DDD
Keywords: left bundle branch block; pacemaker; physiologic stimulation
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: 3D Electroanatomical Mapping (NavX) — To utilize 3D mapping as a tool to explore electro-anatomical and electrocardiographic characteristics of the Left Bundle Branch Area. Patients will undergo placement of standard Left Bundle Area pacing leads for routine indications, during the implantation procedure electro-anatomical map of the target area and neighboring tissues will be created. Map characteristics will be analyzed and used intra-operatively to assist with lead placement along with standard pacing metrics and standard X-ray criteria. We plan on prospectively reviewing the data found from 3D mapping the left bundle branch implantation cases.
  Other Names: Implantation of a standard Left Bundle Area pacing lead and pacing device

SUMMARY:
This study will utilize 3D mapping as a tool to explore electro-anatomical and electrocardiographic characteristics of the Left Bundle Branch Area. We plan on prospectively reviewing the data found from 3D mapping the left bundle branch implantation cases and using the data to improve understanding of electro-anatomical characteristics of this area for a better definition of the implantation target and depth.

DETAILED DESCRIPTION:
This is an observational study that will provide the data for further hypothesis generation and confirmation in a larger study. We will define and record electro-anatomical characteristics of the interventricular septum and surrounding areas. Several electro-anatomical characteristics will be measured during the lead placement into the Left Bundle Branch Area. Mapping will be performed with the pacing lead. We will collect electrocardiographic markers of successful and unsuccessful LBBA pacemaker implantation attempts and correlate them with electro-anatomical information.

ELIGIBILITY:
Inclusion Criteria:

* 30 consecutive patients ages 18 through 88 that undergo Left Bundle Branch area pacemaker implantation.

Exclusion Criteria:

* Recent MI-less than 3 months
* Recent Percutaneous Coronary Revascularization-less than 2 weeks
* Recent Open-Heart Procedures (CABG, Valvular procedures, etc.)-less than 1 month
* Patients who are acutely ill and unstable, from the investigator's perspective, but require an urgent permanent pacemaker

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients ages 18 through 88 that undergo Left Bundle Branch area pacemaker implantation for standard pacemaker indications at one location (Steward St. Elizabeth Medical Center).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Electroanatomical characteristics of the target area for Left Bundle lead implantation | Through study completion, an average of 1 year
  Electroanatomical metrics

CONTACTS AND LOCATIONS:
Overall Officials: Michael Orlov, MD, PhD, Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (1):
- St. Elizabeth's Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Orlov MV, Jahangir A, McKelvey D, Armstrong J, Maslov M, Monin AJ, Koulouridis I, Casavant D, Wylie JV. His bundle pacing insights from electroanatomical mapping: Topography and pacing targets. J Cardiovasc Electrophysiol. 2020 Oct;31(10):2737-2743. doi: 10.1111/jce.14672. Epub 2020 Jul 23. PMID 32666617
- [Result] Orlov MV, Nikolaychuk M, Koulouridis I, Goldman A, Natan S, Armstrong J, Bhattacharya A, Hicks A, King M, Wylie J. Left bundle area pacing: Guiding implant depth by ring measurements. Heart Rhythm. 2023 Jan;20(1):55-60. doi: 10.1016/j.hrthm.2022.09.013. Epub 2022 Sep 21. PMID 36152975
- [Result] Orlov MV, Koulouridis I, Monin AJ, Casavant D, Maslov M, Erez A, Hicks A, Aoun J, Wylie JV. Direct Visualization of the His Bundle Pacing Lead Placement by 3-Dimensional Electroanatomic Mapping: Technique, Anatomy, and Practical Considerations. Circ Arrhythm Electrophysiol. 2019 Feb;12(2):e006801. doi: 10.1161/CIRCEP.118.006801. PMID 30739495